CLINICAL TRIAL: NCT04795882
Title: An Open Label, Phase 1 Study Evaluating the Activity of Modular CAR T for mYeloma
Brief Title: A New Study Evaluating the Activity of Modular CAR T for mYeloma
Acronym: MCARTY
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL 129642
Record Dates: First submitted 2021-03-02; First posted 2021-03-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Rolling 6 trial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: BCMA CAR T cells (Experimental): Treatment with Advanced Therapy Investigational Product (ATIMP): BCMA CAR T-cells
  Interventions: Biological: BCMA CAR T cells
- Cohort 2: BCMA/CD19 CAR T cells (Experimental): Treatment with Advanced Therapy Investigational Product (ATIMP): BCMA/CD19 CAR T-cells
  Interventions: Biological: BCMA/CD19 CAR T cells

INTERVENTIONS:
Biological: BCMA CAR T cells — Infusion with ATIMP: BCMA CAR T-cells
  Arms: Cohort 1: BCMA CAR T cells
Biological: BCMA/CD19 CAR T cells — Infusion with ATIMP: BCMA/CD19 CAR T-cells
  Arms: Cohort 2: BCMA/CD19 CAR T cells

SUMMARY:
This is a Phase 1 rolling 6 trial design evaluating safety of a novel BCMA Chimeric Antigen Receptor (CAR) alone and of CAR T cells engineered to co-express BCMA CAR and a CD19 CAR in patients with relapsed / refractory Multiple Myeloma.

The study will assess the feasibility of generating these Advanced Therapy Investigational Products (ATIMPs) and the safety of administering the CAR T cells (either BCMA alone or co-expressed with CD19) in patients with relapsed / refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a Phase 1 rolling 6 trial design evaluating safety of a novel BCMA CAR alone and of CAR T cells engineered to co-express BCMA CAR and a CD19 CAR in patients with triple refractory Multiple Myeloma.

The first 3-6 patients will be treated at the lower dose of BCMA CAR T cells in cohort 1 (50 x 10^6 cells). If the lower dose is deemed tolerable, recruitment into cohort 1 at a higher dose (150 x 10^6 BCMA CAR T cells) and cohort 2 at a dose of 50 x 10^6 BCMA/CD19 cells will begin in parallel.

* If the 50 x 10^6 cells BCMA/CD19 CAR dose in cohort 2 is deemed intolerable, then no further patients will be recruited to cohort 2.
* If both 150 x 10^6 cells BCMA CAR (cohort 1) and 50 x 10^6 cells BCMA/CD19 CAR (cohort 2) are deemed tolerable then recruitment will begin to a higher BCMA/CD19 CAR dose of 150 x 10^6 cells.
* If 150 x 10^6 cells BCMA CAR is intolerable and 50 x 10^6 cells BCMA/CD19 CAR is tolerable then no further patients will be recruited to cohorts 1 or 2.

With the 150x10^6 cells dose being deemed tolerable in both cohorts 1 and 2, a dose level 3 of 450x10^6 CAR T cells has been added to the design via a substantial amendment. Dose level 3 will first open in cohort 1 and, if deemed tolerable, will then proceed to be opened in cohort 2.

A Summary of dosing on trial is outlined below:

Cohort 1 (BCMA CAR-T cells)

* Dose level 1: 50x10^6 BCMA CAR-T cells
* Dose level 2: 150x10^6 BCMA CAR-T cells
* Dose level 3: 450x10^6 BCMA CAR-T cells administered as a split dose on D0 and D7 (if 1st infusion tolerated well)

Cohort 2 (BCMA/CD19 CAR-T cells)

* Dose level 1: 50x10^6 BCMA/CD19 CAR-T cells
* Dose level 2: 150x10^6 BCMA/CD19 CAR-T cells
* Dose level 3: 450x10^6 BCMA/CD19 CAR-T cells administered as a split dose on D0 and D7 (if 1st infusion tolerated well)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Relapsed/Refractory Multiple Myeloma
3. Secretory disease: PP≥5g/L and/or sFLC≥100mg/L of involved light chain with abnormal K:L ratio.
4. ≥3 prior lines of therapies (including proteasome inhibitor, IMiD, anti CD38 antibody)
5. Refractory to last line of therapy (not achieved at least PR and progressed within 60 days of last dose or achieved at least PR but progressed within 6 months of last dose)
6. Has previously received or is not suitable for ASCT
7. Eastern Cooperative Oncology Group (ECOG) performance status 0/1
8. Creatinine Clearance (CrCl)≥40ml/min, Absolute Neutrophil Count (ANC)≥1x10^9/L, Platelets (plt)≥50x10^9/L, Haemoglobin (Hb)≥80 /L, lymphocyte count ≥0.3x10^9/L
9. Patients must weigh >30 kg
10. Agreement to have a pregnancy test, use adequate contraception (if applicable)
11. Written informed consent

Exclusion Criteria:

1. Previous diagnosis of systemic light chain amyloidosis
2. Prior treatment with investigational or approved gene therapy or cell therapy products
3. Stem cell transplant patients only:

   * allogeneic stem cell transplant within 12 months prior to registration into the study
   * moderate/ severe chronic GVHD (NIH consensus criteria) requiring immunosuppressive therapy and/or systemic steroids
4. Oxygen saturation ≤ 90% on air
5. Patients with clinically significant, uncontrolled heart disease or a recent (within 6 months) cardiac event
6. Left ventricular ejection fraction < 50% (ECHO or MUGA)
7. Corrected QT interval (QTc)>470 ms on ECG
8. Uncontrolled cardiac arrhythmia (patients with rate-controlled atrial fibrillation are not excluded)
9. History or evidence of deep vein thrombosis or pulmonary embolism requiring ongoing therapeutic anticoagulation at preconditioning
10. Chronic renal impairment requiring dialysis
11. Patients with significant liver disease: alanine aminotransferase or aspartate aminotransferase ≥3x upper limit normal (ULN), or total bilirubin ≥25umol/L (1.5mg/dL), except in patients with Gilbert's syndrome, or evidence of end-stage liver disease (e.g. ascites, hepatic encephalopathy)
12. Patients with any major surgical intervention in the last 3 months, cement augmentation for vertebral collapse is permitted
13. Patients with active gastrointestinal bleeding
14. Patients with active infectious bacterial or viral disease requiring treatment
15. Known active central nervous system involvement of MM. History or presence of clinically relevant central nervous system pathology such as epilepsy, paresis, aphasia, stroke within 3 months prior to enrolment, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, uncontrolled mental illness, or psychosis
16. Patients receiving corticosteroids at a dose of >5 mg prednisolone per day (or equivalent) that cannot be discontinued
17. Active autoimmune disease requiring immunosuppression
18. Past or current history of other neoplasms
19. Received any radiotherapy within the last 7 days prior to lymphodepletion or leukapheresis. Localised radiation to a single site, e.g. for bone pain is permitted at any time
20. Patients with any anti-myeloma therapy within the last 7 days prior to LD or leukapheresis
21. Inability to tolerate leucapheresis
22. Life expectancy <3 months
23. Women who are pregnant or breastfeeding
24. Known allergy to albumin or DMSO

Exclusion criteria for CAR-T cell infusion:

1. Active infection requiring systemic anti-microbial therapy, or with temperature more or equal to 38 C within 48 hours before scheduled CAR-T cell infusion
2. Requirement for supplementary oxygen at the time of scheduled CAR-T cell infusion
3. Clinical deterioration of organ functions (hepatic or renal function) exceeding criteria set at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity evaluated by the incidence of grade 3-5 toxicity causally related to the Advanced Therapy Investigational Product (ATIMP) | 28 days
  The incidence of grade 3-5 toxicity assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and the American Society for Transplantation and Cellular Therapy (ASTCT) Cytokine Release Syndrome (CRS) and Neurotoxicity tool
Feasibility of manufacturing CAR T-cells evaluated by the number of therapeutic products generated | 30 days
  Feasibility of generation of CAR T cells as evaluated by the number of therapeutic products generated.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, County (Optional), United Kingdom

IPD SHARING:
Plan to Share IPD: No